CLINICAL TRIAL: NCT00458575
Title: A Phase I Open Label Non-comparative Study Evaluating the Safety of a Single, Unilateral, Subretinal Administration of CNTO 2476 in Advanced Retinitis Pigmentosa
Brief Title: A Study to Evaluate the Safety of CNTO 2476 in Patients With Advanced Retinitis Pigmentosa
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Internal Business Decision
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR013210; CNTO2476RPG1001 (Other: Centocor, Inc)
Record Dates: First submitted 2007-04-10; First posted 2007-04-11 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Retinitis Pigmentosa
Keywords: Retinitis Pigmentosa; Advanced retinitis pigmentosa (RP); CNTO 2476; Subretinal; Human umbilical tissue-derived cells (hUTC); Light perception (LP); Hand motion (HM)
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CNTO 2476 (Experimental): Participants 1 to 4: advanced retinitis pigmentosa (RP) with light perception only (LP); Participant 5: combination visual acuity of LP in the treated eye and no better than hand motion (HM) in the fellow eye; and Participants 6 to 9: advanced RP with hand motion (HM) will receive different dose levels of CNTO 2476.
  Interventions: Drug: CNTO 2476

INTERVENTIONS:
Drug: CNTO 2476 — Participant 1 will receive 5.6x100000; Participants 2, 3, 5, 6, and 7 will receive 6.0x10000; Participant 4 will receive 3.0x100000; and Participants 8 and 9 will receive 1.2x100000 of CNTO 2476 as a single dose of viable cells in phosphate buffered saline (PBS) in a total volume of 100 μL injected subretinally.

SUMMARY:
The main purpose of this study is to evaluate the preliminary safety and immunogenicity (ability of an antigen to provoke immune response in the human body) of CNTO 2476, administered subretinally, in participants with advanced retinitis pigmentosa (RP; disease of the eye that leads to loss of vision and blindness) with either light perception only (LP) or hand motion (HM).

DETAILED DESCRIPTION:
The study will be an open-label (all people know the identity of the intervention), first in human safety study. Nine adult men and women with advanced RP with LP only (first 5 participants) or not better than HM bilaterally (subsequent 4 participants) in both eyes will be enrolled. Participant 5 may have combination visual acuity of LP in the treated eye and no better than HM in the fellow eye. Treatment will proceed on a cohort basis ie, Cohort I: Participant 1; Cohort II: Participant 2; Cohort III: Participant 3 and 4; Cohort IV: Participant 5, 6, and 7; and Cohort V: Participant 8 and 9. The initial participants for each cohort must have completed at least 4 weeks of post-treatment follow-up before participants in the next cohort may be treated. There are 2 safety assessment phases in this study: the main phase approximately 12 months from the time the participant is eligible to enter the study and the long-term safety follow-up phase of 4 additional years. The total length of the participation in the study could last up to 5 years (including both the main and safety follow-up phases).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of retinitis pigmentosa that is not part of another systemic disease
* Vision deficit characterized by vision that is not better than either light perception (Group 1) or hand motion (Group 2) in both eyes
* Normal hematology and chemistry lab results
* Participant is suitable candidate for ophthalmologic surgery

Exclusion Criteria:

* Other significant ophthalmologic diseases or any other ophthalmologic condition that interferes with ophthalmologic examination
* Women of childbearing potential
* Ocular hypertension
* Other serious medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Number of adverse events as a measure of safety and tolerability | Up to 5 years from the time participant is eligible to enter study
Level of anti-CNTO 2476 antibody in blood for immunogenicity testing | Baseline, Days 7 and 15, Weeks 3 and 4, Months 2, 3, 6, 12, 24, 36, 48, and 60

SECONDARY OUTCOMES:
Change from baseline in retinal structure and visual function | Up to 5 years from the time participant is eligible to enter study
  This will be assessed by optical coherence tomography (OCT), fluorescein angiography (FA), fundus photography, and visual field sensitivity (FFST).

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.
Locations (3):
- United States (3):
  - Miami, Florida
  - Southwest Portland, Oregon
  - Dallas, Texas

REFERENCES:
- [Derived] Davis JL. The Blunt End: Surgical Challenges of Gene Therapy for Inherited Retinal Diseases. Am J Ophthalmol. 2018 Dec;196:xxv-xxix. doi: 10.1016/j.ajo.2018.08.038. Epub 2018 Sep 5. PMID 30194931